CLINICAL TRIAL: NCT02578667
Title: Gorbly Compression Device for Use in Image-guided Procedures
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: study cancelled
Sponsor: University of Miami (Other)
Collaborators: Wallace H Coulter Center for Translational Research (Other)
Responsible Party: Principal Investigator, Issam Kably, Assistant Professor, University of Miami
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 20150294
Record Dates: First submitted 2015-10-07; First posted 2015-10-19 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Neoplasm; Sepsis
MeSH Terms: conditions — Neoplasms; Sepsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gorbly Compression not needed (No Intervention)
- Gorbly Compression may benefit (Experimental): the use of the Gorbly device with the consent of the patient
  Interventions: Device: Gorbly Compression Device

INTERVENTIONS:
Device: Gorbly Compression Device — The compression device provides a way to displace critical structures along the path from skin to target, retract excess body wall tissue, and provide mechanical stabilization in a repeatable and sustainable fashion.
  Arms: Gorbly Compression may benefit

SUMMARY:
Prospective cohort study. All patients presenting for percutaneous abdomino-pelvic soft tissue ablation, biopsy, or drainage performed under the care of Dr. Issam Kably will become part of the study population. Based on prior imaging and/or imaging at the time of the procedure, patients will fall into two groups, those for whom no compression is necessary to complete the procedure and those for whom compression may provide benefit. These would be selected based on Dr. Kably's experience as a practicing academic, fellowship-trained, and CAQ'ed interventional radiologist. The latter group would then further subdivide into those who give consent for use of the compression device and those who do not consent. Results of each group would be measured including the following: termination versus successful completion of the procedure; adverse events including bleeding or damage to surrounding structures necessitating further medical or surgical intervention.

ELIGIBILITY:
Inclusion Criteria:

* All-comers presenting for percutaneous abdomino-pelvic soft tissue ablation, biopsy, or drainage .

Exclusion Criteria:

* Open surgical or traumatic abdominal wall.
* Active abdominal wall infection.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-12; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
The percentage of procedures (i.e., ablations, biopsies, or drainages) that are allowed successful completion. | intraoperative

SECONDARY OUTCOMES:
The rate of complication of bleeding or damage to the surrounding vessels or organs by use of the compression device. | intraoperative

CONTACTS AND LOCATIONS:
Overall Officials: Issam Kably, MD, Principal Investigator — University of Miami
Locations (1):
- Jackson Memorial Hospital, Miami, Florida, United States